CLINICAL TRIAL: NCT01758471
Title: An Open-label, Randomized , Phase 4 Study to Compare the Different Efficacies of α-glucosidase Inhibitor and Sulfonylurea on Improvement of Intestinal Microbiome and Serum Incretins in Patients With Type 2 Diabetes
Brief Title: Efficacy of Acarbose on Intestinal Microbiome and Incretins of Type 2 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Guang Ning, Vice president of Ruijin Hospital affiliated to Shanghai Jiao Tong University School of Medicine, Director of Shanghai Institute for Endocrine and Metabolic Diseases, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CCEMD017
Record Dates: First submitted 2012-12-24; First posted 2013-01-01 (Estimated); Last update posted 2013-01-01 (Estimated); Status verified 2012-12

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; gut microbiome; incretin; Sulfonylurea; α-glucosidase inhibitor
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glipizide; Acarbose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acarbose (Experimental): The minimum dosage of acarbose in this study is 100mg tid p.o.(oral) for 3 month. With this dosage, patients should have similar glycemic control with those using glipizide, that is FBG(fasting blood glucose)<7.0,PBG(postprandial blood glucose)<10.0
  Interventions: Drug: Acarbose
- glipizide (Active Comparator): There is no fixed dosage of glipizide to control hyperglycemia for patients in this group. As long as the targeted blood glucose concentration is reached, FBG< 7.0, PBG< 10.0, patients will have the least dosage of glipizide according to their glucose level.
  Interventions: Drug: Glipizide

INTERVENTIONS:
Drug: Glipizide — glipizide 5mg per pill 5mg tid p.o. for 3 month
  Arms: glipizide
Drug: Acarbose — Acarbose 50mg per pill 100mg to 150mgtid p.o.（oral） for 3 month
  Other Names: glucobay
  Arms: Acarbose

SUMMARY:
This study is aimed to investigate the effect of acarbose on intestinal microbiome and incretins, therefore to explore the new pathways or new targets to treat type 2 diabetes.

DETAILED DESCRIPTION:
In recent years, Endocrinologist and Diabetologists have found that intestine might serve as a novel target for treating diabetes or other metabolic diseases. Incretins are well-known hormones secreted from intestine, such as CCK（Cholecystokinin), Serotonin, GIP(gastric inhibitory polypeptide) and GLP-1(glucagon like peptide 1), to help control wholesome metabolic status through their effects on pancreatic islet cells, hypothalamus neurons and gastrointestinal movement. Gut microbiome has been recently revealed exerting major effect on host's immune system and metabolic balance with its various metabolites and components.

α-glucosidase inhibitors have been used as anti-diabetes medicine for dozens of years. They are known to be effective by delaying glucose absorption in small intestine. Questions then have been arisen that if delaying glucose absorption changes the intestinal bacteria flora component by increasing bacteria fed on glucose, or that if it influences incretin secretion, since most glucose sensitive L cell (secreting GLP-1) were located in the distal part of small intestine and colon, and that if the hypoglycemia effect of α-glucosidase inhibitors might be mediated by either intestinal flora or incretins.

To address the questions above and to find the new targets from the intestine to treat diabetes, we therefore design this study, taking advantage of clinical trial and basic biomedical studies to find if α-glucosidase inhibitor- Acarbose (Bayer, Corp.) could change the profile of intestinal incretins and microbiome.

Study design:

1. Multi-center, open label, randomized, positive control cohort.
2. 110 cases of newly-diagnosed Type-2 Diabetes patients from five clinic centers from Shanghai, China Mainland.
3. All patients will sign the consent and screened by the criteria before enrolled by this study.
4. 55 cases of Type 2 Diabetes will be assigned to glucobay treatment and another 55 will take glipizide.
5. 50 healthy volunteers for baseline data comparison.
6. The duration of whole study will be 3 month.

   1. Before treatment, all the patients will be required to have OGTT(oral glucose tolerant test) and IRT(insulin release test) test and give their feces. Standard meals will be required one day before the feces are collected.
   2. In 3 months, all patients will take the medicine and their glucose will be monitored closely by visiting outpatient office once a month.
   3. In the end of the study, patients will be required to receive OGTT and IRT and give their feces again.
7. Serum and feces will be stored at -80℃ for further biomarkers investigation and microbiome sequencing.
8. After 3 months intervention, patients will be observed for another 3 month with access to routine clinic visiting.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed Type 2 Diabetes, without any previous drug treatment,
* 7.0 mmol/l <=FBG<=13.O mmol/l, HbA1C <=10%
* Body mass index (BMI) < 35kg/m2 (inclusive);
* Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures are conducted
* Having good study compliance

Exclusion Criteria:

* Intestinal surgery or recent abdominal surgery within 1 year
* Taken immunosuppressive agents, steroid,antidiarrhea agents, antibiotics and other gastrointestinal motility agents within 3 months
* Severe liver dysfunction, including serum alanine aminotransferase concentration more than 2.5 times above upper limit of normal range, abnormal renal function (GFR < 60ml/min)
* Other severe conditions which will put the patients in high risk during the study
* Any clinically significant allergic disease
* Women in pregnancy or under breast feeding

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
euglycemia | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Guang Ning, M.D. Ph.D., Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Clinic Center for Endocrine and Metabolic Diseases, Ruijin Hospital, Shanghai Institute for Endocrine and Metabolic Diseases, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Ni M, Chen Y, Gu W, Zhang Y, Xu M, Gu Y, Chen Y, Zhu Y, Wang X, Luo Y, Xu Y, Lin X, Zeng YA, Liu R, Wang J. Association Between Circulating Gremlin 2 and beta-Cell Function Among Participants With Prediabetes and Type 2 Diabetes. J Diabetes. 2025 Apr;17(4):e70090. doi: 10.1111/1753-0407.70090. PMID 40270326